CLINICAL TRIAL: NCT03510013
Title: 1-1-8 Wash-in for Sevoflurane Low Flow Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE601228
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia
Keywords: low flow anesthesia; wash-in; sevoflurane
MeSH Terms: interventions — Sevoflurane; Anesthetics, Inhalation

STUDY DESIGN:
Intervention Model Description: All participants will receive sevoflurane 8% with O2:N2O or O2:air 1:1 L/min under controlled ventilation. Time to achieve alveolar concentration of sevoflurane of 1%, 1.5%, 2%, 2.5%, 3% and 3.5% will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1-1-8 wash-in (Experimental): Wash-in using O2:N2O or O2:air 1:1 L/min with sevoflurane 8%
  Interventions: Procedure: 1-1-8 wash-in; Drug: Sevoflurane

INTERVENTIONS:
Procedure: 1-1-8 wash-in — wash-in phase during start of low flow anesthesia
Drug: Sevoflurane — Drug used for wash-in protocol
  Other Names: Inhalation anesthetic

SUMMARY:
The investigators propose a new wash-in technique for sevoflurane low flow anesthesia with fresh gas flow of O2:N2O or O2:air 1:1 L/min with sevoflurane 8%.

The objective of this study is to identify time to achieve alveolar concentration of sevoflurane at 1, 1.5, 2, 2.5, 3, and 3.5%

DETAILED DESCRIPTION:
The benefits of low flow anesthesia are economic, less pollution, more heat and humidity preservation but it requires appropriate wash-in phase. The current wash-in protocols for sevoflurane are complicated and time consuming. The investigators propose a new 1-1-8 sevoflurane wash-in protocol which is more simple and predictable.

The objective of this study is to identify time to achieve alveolar concentration of sevoflurane at 1, 1.5, 2, 2.5, 3, and 3.5% with 1-1-8 wash-in protocol.

All patients will receive iv propofol 2 mg/kg as induction agent and succinyl choline 1.5 mg/kg for intubation. Then the ventilation will be controlled to achieve end-tidal CO2 30-35 mmHg with O2:N2O or O2:air 1:1 L/min with sevoflurane 8%. Time to achieve alveolar concentration of sevoflurane at 1, 1.5, 2, 2.5, 3, and 3.5% will be recorded and analyzed. After that, the concentration of sevoflurane and anesthetic technique will be adjusted to requirement of anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-II
* age 18-65 years

Exclusion Criteria:

* BMI > 35
* contraindicated for N2O
* • with pulmonary or cardiac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Time | participants will be followed until alveolar concentration of sevoflurane reaches 3.5%, as expected of 10 minutes
  Time (in second) to achieve alveolar concentration of sevoflurane 1, 1.5, 2, 2.5, 3, and 3.5%

SECONDARY OUTCOMES:
Heart rate | participants will be followed until alveolar concentration of sevoflurane reaches 3.5%, as expected of 10 minutes]
  Heart rate (beat/min) at alveolar concentration of sevoflurane of 1, 1.5, 2, 2.5, 3 and 3.5%
Blood pressure | participants will be followed until alveolar concentration of sevoflurane reaches 3.5%, as expected of 10 minutes]
  Blood pressure (systolic and diastolic (mmHg)) at alveolar concentration of sevoflurane of 1, 1.5, 2, 2.5, 3 and 3.5%

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tribuddharat S, Sathitkarnmanee T, Vattanasiriporn N, Thananun M, Nonlhaopol D, Somdee W. 1-1-8 one-step sevoflurane wash-in scheme for low-flow anesthesia: simple, rapid, and predictable induction. BMC Anesthesiol. 2020 Jan 24;20(1):23. doi: 10.1186/s12871-020-0940-2. PMID 31980020